CLINICAL TRIAL: NCT04592809
Title: Double-Blind Randomized Controlled Trial of Acute-Course of Ketamine Versus Midazolam for Recurrence of Suicidality in Adolescents
Brief Title: Ketamine Versus Midazolam for Recurrence of Suicidality in Adolescents
Acronym: TASK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Madhukar H. Trivedi, MD, Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU-2020-0973; R01MH125181 (NIH)
Record Dates: First submitted 2020-09-29; First posted 2020-10-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Suicide, Attempted; Suicide and Depression; Suicide Threat
Keywords: depression; adolescent; suicidal ideation; suicide attempt; teen; child; intensive outpatient; inpatient hospitalization; depression treatment; suicide treatment
MeSH Terms: conditions — Suicide, Attempted; Suicide; Depression; Suicidal Ideation | interventions — Ketamine; Midazolam

STUDY DESIGN:
Intervention Model Description: Youth will be randomized in 1:1 fashion to either intravenous ketamine (0.5 mg/kg) or midazolam (0.02 mg/kg) twice weekly for 2 weeks followed by weekly visits for 10 weeks (for a total of 12-week post-randomization observation period).
Who Masked: Participant, Care Provider, Investigator
Masking Description: The investigator, patient, and study staff will be blinded. Packaging and labeling of the study drugs will be performed by the research pharmacy in a way to ensure blinding throughout the study.
  No members of the study team will have access to the randomization scheme during the conduct of the study. The Research Pharmacist and the CDRC (Center for Depression Research and Clinical Care) Program Manager will have access to the treatment assignment in the event of an emergency. The treatment code must not be broken except in medical emergencies when the appropriate management of the patient necessitates knowledge of the treatment randomization. The investigator retains the right to break the code for serious adverse events (SAEs) that are unexpected and are suspected to be causally related to a study drug and that potentially require expedited reporting to regulatory authorities.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ketamine (Active Comparator): 0.5 mg/kg intravenous ketamine will be administered 4 times in a 2 week period. Ketamine will be dissolved in 0.9% sodium chloride in a total volume of 100ml and administered with a syringe infusion pump at a constant rate.
  Interventions: Drug: Ketamine Hydrochloride; Drug: Midazolam Hydrochloride
- Midazolam (Active Comparator): 0.02 mg/kg midazolam will be administered 4 times in a 2 week period. Midazolam will be dissolved in 0.9% sodium chloride in a total volume of 100ml and administered with a syringe infusion pump at a constant rate.
  Interventions: Drug: Ketamine Hydrochloride; Drug: Midazolam Hydrochloride

INTERVENTIONS:
Drug: Ketamine Hydrochloride — infused over a 40 minute period
  Other Names: Ketalar
Drug: Midazolam Hydrochloride — infused over a 40 minute period
  Other Names: Versed

SUMMARY:
This project aims to examine the signal of efficacy of ketamine, a rapidly acting medication shown to decrease suicidality in adults in as short as hours or days, as opposed to weeks.

The study design is a double-blind, randomized, active-control trial of adolescents (ages 13-18 years) with recent suicidal behaviors (suicide attempt or increased suicidal ideation). All participants must be receiving standard of care treatment which may range broadly from both outpatient and inpatient programs which include clinically indicated psychosocial and/or psychopharmacological treatments. Ketamine/midazolam treatment will occur twice weekly during the first two weeks of the study, followed by weekly assessments through week 12.

DETAILED DESCRIPTION:
Adolescent patients (ages 13-18) who have recent suicidality (defined as suicide attempt or urgent evaluation for a suicidal ideation or behavior), and who are receiving standard of care treatment (e.g., psychosocial and/or psychopharmacological treatment) will be recruited for participation in the study. Upon informed consent/assent, screening data will be collected regarding mood symptoms, suicidal ideation and behavior, associated comorbidities, and treatment history. Youth participants will be randomized to receive infusions of either ketamine or midazolam, which will be provided twice weekly for two weeks. Participants will then have follow-up assessments visits through week 12 to continue to monitoring outcome measures.

Participants may be recruited directly from their standard care outpatient provider, SPARC Intensive Outpatient Program (IOP) located at Children's Health Medical Center, from the Children's Health Emergency Department (ED) or inpatient psychiatric unit located at the Dallas campus. Participants may also be recruited into the study even if they are seen in the in emergency departments or inpatient hospitalization outside of University of Texas (UT) Southwestern and Children's Health Medical Center. Recruitment and consent procedures may begin during ED or inpatient hospitalization; however, as the study is an outpatient study, study procedures will not begin until the participant is discharged from the ED or inpatient hospital.

Recruitment efforts will target medically healthy male and female youths with recent suicide events who are either seeking care at an emergency room, admitted to an inpatient unit, enrolled in an IOP, or receiving adequate outpatient care with either psychopharmacological or psychosocial treatment following a suicide event.

Enrollment of 114 subjects is expected to take place over a period of approximately 36 months. Enrolled participants will be involved in the study for approximately 14 weeks. Visits include a Screening Visit, 4 Study Intervention Visits, and 11 Follow-Up Visits (combination of in-person and remote visits). Multiple streams of outcome measures will be utilized for this protocol, including self-report measures, research assessor-completed measures, clinic level measures, and behavioral measures.

Aim 1. Evaluate reduction in repeat suicidal events with ketamine.

Aim 2. Evaluate reduction in implicit suicidal cognition with ketamine.

Aim 3. Evaluate reduction in depressive symptoms and suicidality with ketamine.

ELIGIBILITY:
Inclusion Criteria

Study participants must:

1. Be adolescents (aged 13-18 years);
2. Have had a recent suicidal event (suicide attempt or significant suicidal ideation with a plan or intent warranting emergency evaluation or inpatient hospitalization within the past 90 days);
3. Receiving standard of care treatment that includes clinically indicated psychosocial and/or psychopharmacological treatment;
4. Have a current primary diagnosis of a depressive disorder based on the MINI-KID (other psychiatric disorders are acceptable, but must not be primary);
5. Participants must be able to complete assessments in English. However, the parent(s) or legal guardians of minors may either speak English or Spanish
6. Use effective method of contraception during and for 90 days following the end of treatment for female and male participants. Recommended methods of birth control are namely, consistent use of an approved hormonal birth control (pill/patches, rings), an intrauterine device (IUD), contraceptive injection, double barrier methods, sexual abstinence, or sterilization;

Exclusion Criteria

Study participants must not:

1. Have a psychotic disorder, such as lifetime schizophrenia, or a pervasive or intellectual developmental disorder requiring substantial or very substantial support;
2. Have current mania, hypomania, mixed episode, or obsessive-compulsive disorder;
3. Have a primary diagnosis other than a depressive disorder;
4. Have moderate to severe alcohol or substance use disorder within the past six months (based on MINI-KID); If there is a positive urine drug screen at screening, the urine drug screen will be repeated at each infusion visit. Positive urine drug screen will be reviewed by study physician and infusion will proceed as long as no safety risk was identified;
5. If female, be pregnant, lactating, or nursing; Women of childbearing potential must have a negative urine pregnancy test prior to all infusions;
6. Have unstable medical conditions (stable for less than 3 months) or with clinically significant laboratory values or an electrocardiogram (ECG) that would pose significant risk;
7. Be at serious suicidal risk that cannot be managed in the outpatient setting;
8. Have prior treatment for depression with or contraindications to ketamine, esketamine, or, midazolam;
9. Treatment with medications that may alter pharmacokinetics of ketamine, including moderate-to-strong inhibitors or inducers of CYP3A4 and CYP2B6, is exclusionary. Regarding pharmacodynamic interactions, medications that may increase heart rate or blood pressure such as the ADHD stimulant medications will be permitted with last dose at least 24 hours prior to infusion. All concomitant medications will be evaluated by the study physician to determine if the type and dose of concomitant medication requires discontinuation and will be excluded if the concomitant medication could substantially increase the risk of study infusion. A complete list of medications that are Not Allowed is available in Appendix D of the protocol. The study team will not ask the participant to discontinue any treatment (except for not taking ADHD medications for 24 hours before study treatment) just for the sake of taking part in this study;
10. Weigh >120 kilograms at baseline. If participants are enrolled but exceed 120 kilograms at any time during the treatment period, they will be removed from the treatment portion of the study.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
The primary outcome for the study is "suicidal events". Suicidal event is defined as a suicide attempt, or emergency department visit or inpatient hospitalization due to suicidality. | 12 weeks
  Concise Health Risk Tracking Clinician-Rated Behavior Module (CHRT-C) will be used to identify suicidal events. The CHRT-C consists of nine clinician-rated yes/no items about specific behaviors (i.e., suicidal ideation, suicidal attempt, preparatory acts, non-suicidal self-injury (NSSI), other injuries, etc.). At the initial administration, this instrument captures lifetime information; at subsequent administrations, it will capture information since the last visit.

SECONDARY OUTCOMES:
Death/Suicide Implicit Association Test (IAT) | 2 weeks
  The IAT is a performance-based measure of cognition that has demonstrated good reliability and sensitivity to change. The IAT measures associations based on response latency where the response time is compared across categorization tasks.
Depression symptoms as measured by CHRT-SR a self report measure | 2 weeks
  (specify for each) Concise Health Risk Tracking Self-Report (CHRT-SR) consists of 14 questions with responses ranging from 0 (strongly disagree) to 4 (strongly agree). 1) the Propensity subscale, which consists of 9 questions and 4 factors (pessimism, helplessness, social support, and despair) and a score range of 0-36; and the Suicidal Thoughts subscale, which consists of 3 questions and a score range of 0-9 (which will serve as the primary suicidal behavior outcome in this study); and 3) Impulsivity, which consists of 2 questions and a score range of 0-6. A total score is also calculated, ranging from 0 to 56.
Number of participants with suicidal events/behaviors as measured by CHRT-C a self report measure | 2 week
  Concise Health Risk Tracking Clinician-Rated Behavior Module (CHRT-C). consists of nine clinician-rated yes/no items about specific behaviors (i.e., suicidal ideation, suicidal attempt, preparatory acts, non-suicidal self-injury (NSSI), other injuries, etc.). At the initial administration, this instrument captures lifetime information; at subsequent administrations, it will capture information since the last visit. a yes on any of the 9 questions indicates presence of suicidal event/behaviors (ideation, attempt, preparatory acts, non suicidal self injury, other injury).
Depression symptoms as measured by the Inventory of Depressive Symptomatology (IDS), self-report measure | 2 weeks
  The Inventory of Depressive Symptomatology (IDS) Self Report is a depressive symptom severity measure that rates all nine criterion symptoms of MDD, and includes an irritability item for adolescents. The self report (IDS-SR) will be completed at each visit.

CONTACTS AND LOCATIONS:
Overall Officials: Madhukar Trivedi, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No